CLINICAL TRIAL: NCT05117086
Title: DASH Diet in Heart Failure Pilot Study - Integration and Effectiveness of Medical Nutrition Therapy Counseling on DASH Diet in the Management of Heart Failure Patients in an Academic Outpatient Cardiology Clinic
Brief Title: DASH Diet in Heart Failure Outpatients
Acronym: DASH-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: American College of Cardiology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1770356
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Intervention Model Description: Single arm pragmatic trial with pre- and post- assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Intervention Arm (Experimental): Subjects will receive the active intervention of nutrition education and medical nutrition therapy counseling for dietary and behavioral lifestyle changes. The focus will be on DASH diet implementation and adherence for management of heart failure. The subjects will have 4 study visits with a Registered Dietitian over 6 months (visits at 1, 2, 3, and 6 months). Outcome measures will be assessed at baseline, 3 and 6 months.
  Interventions: Behavioral: DASH diet

INTERVENTIONS:
Behavioral: DASH diet — Nutrition education and counseling on DASH diet, behavioral and lifestyle modifications

SUMMARY:
The purpose of this study is to refine the classification of the effectiveness of the DASH diet for outpatient heart failure (HF) management, using behavioral, clinical, and laboratory correlative science approaches.

DETAILED DESCRIPTION:
The overall objective of this pilot study is to refine the classification of the effectiveness of the DASH diet for outpatient HF management using behavioral, clinical, and laboratory correlative science approaches. The investigators will integrate the use and evaluation of DASH diet nutrition education in a clinical population using a pragmatic study approach. The investigators will assess dietary behavior change. The investigators will assess the medical effectiveness of the DASH diet to improve patient symptomology and clinical biomarkers. Exploratory investigations will involve metabolomics analyses of plasma samples for biomarker discovery of clinical phenotypes in HF patients, to characterize metabolic profiles related to dietary exposure.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure diagnosis
* Guideline directed medical therapy optimization on stable regimen at least 30 days

Exclusion Criteria:

* BMI < 18/5 kg/m squared
* cardiac cachexia
* end-stage renal disease or dialysis
* acute inflammatory condition
* uncontrolled arrhythmias or ischemia
* status post heart transplant or implanted left ventricular assist device

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-06-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dietary intake | Dietary intake at baseline
  Dietary intake assessed by nutrient analysis of food records
Dietary intake | Dietary intake at 3 months
  Dietary intake assessed by nutrient analysis of food records
Dietary intake | Dietary intake at 6 months
  Dietary intake assessed by nutrient analysis of food records
Diet score | Dietary intake at baseline
  Dietary intake assessed by calculation of DASH diet score (Dietary Approaches to Stop Hypertension diet score). Minimum to Maximum values: 8-40 Higher scores mean better outcome and diet composition.
Diet score | Dietary intake at 3 months
  Dietary intake assessed by calculation of DASH diet score (Dietary Approaches to Stop Hypertension diet score). Minimum to Maximum values: 8-40 Higher scores mean better outcome and diet composition.
Diet score | Dietary intake at 6 months
  Dietary intake assessed by calculation of DASH diet score (Dietary Approaches to Stop Hypertension diet score). Minimum to Maximum values: 8-40 Higher scores mean better outcome and diet composition.
Blood Pressure | Systolic and diastolic Blood Pressure at baseline
  Blood Pressure assessed with systolic and diastolic pressure
Blood Pressure | Systolic and diastolic Blood Pressure at 3 months
  Blood Pressure assessed with systolic and diastolic pressure
Blood Pressure | Systolic and diastolic Blood Pressure at 6 months
  Blood Pressure assessed with systolic and diastolic pressure

SECONDARY OUTCOMES:
Heart Failure clinical marker | proBNP at baseline
  proBNP will be assessed as a marker of severity of heart failure
Heart Failure clinical marker | proBNP at 3 months
  proBNP will be assessed as a marker of severity of heart failure
Heart Failure clinical marker | proBNP at 6 months
  proBNP will be assessed as a marker of severity of heart failure
Patient report of HF symptoms | KCCQ at baseline
  Kansas City Cardiomyopathy Questionnaire (KCCQ) will assess patient report of symptoms. Minimum to Maximum values: 0-100. Higher scores represent better outcome.
Patient report of HF symptoms | KCCQ at 3 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ) will assess patient report of symptoms. Minimum to Maximum values: 0-100. Higher scores represent better outcome.
Patient report of HF symptoms | KCCQ at 6 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ) will assess patient report of symptoms. Minimum to Maximum values: 0-100. Higher scores represent better outcome.
Patient report of eating habit self efficacy | Eating Habits at Baseline
  Eating Habits Questionnaire will assess patient report of self efficacy for behavior change around DASH diet eating habits. Minimum to Maximum values:27-135. Higher value is better outcome.
Patient report of eating habit self efficacy | Eating Habits at 3 months
  Eating Habits Questionnaire will assess patient report of self efficacy for behavior change around DASH diet eating habits. Minimum to Maximum values:27-135. Higher value is better outcome.
Patient report of eating habit self efficacy | Eating Habits at 6 months
  Eating Habits Questionnaire will assess patient report of self efficacy for behavior change around DASH diet eating habits. Minimum to Maximum values:27-135. Higher value is better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Francene Steinberg, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Health Center - Cardiology Department, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No